CLINICAL TRIAL: NCT02216162
Title: PROACTIVE Study Evaluation of the Impact of a Multidimensional Geriatric Intervention Program Including a Regular Physical Training, a Medical and Nutritional Follow-up, on Adjuvant Hormonal Treatment Compliance in Breast Cancer Patients Over 70 Years.
Brief Title: PROACTIVE Study Evaluation of the Impact of a Multidimensional Geriatric Intervention Program
Acronym: PROACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-777
Record Dates: First submitted 2014-08-06; First posted 2014-08-13 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
Keywords: oncogeriatrics; adjuvant endocrine therapy; compliance; elderly; Taï Chi; Physical training
MeSH Terms: conditions — Breast Neoplasms; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A: Interventional adapted physical activity + enhanced geriatr (Experimental): Geriatric (functionality, gait, nutrition) follow-up, biological tests, anti-aromatase agents blood dosing, clinical assessment. Weekly Taï-Chi exercises.
  Interventions: Other: Arm A: adapted physical activity + enhanced geriatric follow-up
- Arm B: control (Other): Clinical follow-up according to the Guidelines, annual geriatric and nutritional assessment
  Interventions: Other: No intervention

INTERVENTIONS:
Other: Arm A: adapted physical activity + enhanced geriatric follow-up — Patients have 3-monthly geriatric follow-up with biological tests, anti-aromatase agents blood dosing and a clinical assessment (M3 to M9, M15 to M22 and M27 to M33). Musculoskeletal adverse events and quality of life level will be reported and analgesic treatment adapted. Patients will be proposed weekly Taï-Chi exercises to improve joint flexibility, muscular tonus and balance and reduce fall risk.
  A broader geriatric assessment including functionality, gait analysis and nutrition will be performed each year (M12, M24 and M36).
  Arms: A: Interventional adapted physical activity + enhanced geriatr
Other: No intervention — Usual clinical follow-up
  Arms: Arm B: control

SUMMARY:
PROACTIVE randomized study to evaluate the impact of a multidimensional geriatric intervention on treatment compliance, measured regularly by blood dosing of drug metabolites.

Patients in the intervention group will be proposed:

* A regular geriatric follow up including an attentive screening of joint symptoms and functionality,
* An adapted treatment of join pain,
* Weekly sessions of adapted physical activity (Taï Chi),
* And a systematic correction of vitamin D deficits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 70 years old
* Non metastatic breast cancer, with or without node metastases
* Hormone Receptor (HR) positive breast cancer patients
* Women with breast adenocarcinoma, confirmed by a pathologist and who underwent surgery or radiotherapy
* Introduce an hormonal therapy during 5 years
* Life expectancy > 6 months (at the discretion of the investigator)
* Covered by a Health System where applicable, and/or in compliance with the recommendations of the national laws in force relating to biomedical research
* Patient must be available for follow-up
* Having given written informed consent prior to any procedure related to the study

Exclusion Criteria:

* No other primary malignant tumor < 5-years old except cured in situ cancer of the cervix, in situ urothelial cancer, or basocellular cancer
* Patient with an experimental treatment in the 30 days prior to the enrollment
* Evidence of metastatic disease
* Not under any administrative or legal supervision

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-04-11 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Compliance of an adjuvant hormonal therapy | 3 years of follow up
  Compliance rate is defined as the rate of blood samplings of anti-hormone metabolites in the therapeutic range, within the 7 blood samplings distributed in the 3 years of follow-up

SECONDARY OUTCOMES:
Intensity and duration of musculoskeletal adverse events | 3 years of follow up
  Musculoskeletal adverse events will be graded using NCI CTC version 4.0
Activities of daily living, functional walking capacity and changes in balance | 3 years of follow up
Quality of life | 3 years of follow up
  Using the Functional Assessment of Cancer Therapy General (FACT-G7) questionnaire
Nutritional status | 3 years of follow up
  Using Mini Nutritional Assessment, weight, weight loss, albuminemia
Analgesics consumption | 3 years of follow up
  issued from the exhaustive list of documented concomitant medications

CONTACTS AND LOCATIONS:
Overall Officials: Claire Falandry, MD-PhD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Claire Falandry, Lyon, France